CLINICAL TRIAL: NCT02844088
Title: Evaluation of the Persistence in 2016 of Vaccinal Immunity Against Meningococcus C Among Children and Teenagers Who Received Meningococcus C Conjugate Vaccine in January 2002 During the Puy-de-Dôme Campaign and of Natural Immunity Among Unvaccinated People
Brief Title: Evaluation of Vaccinal and Natural Immunity Against Meningococcus C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-0273; 2015-A01437-42 (Other: 2015-A01437-42)
Record Dates: First submitted 2016-07-12; First posted 2016-07-26 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Prevention of Meningococcus C Infections
Keywords: meningococcus C

ARMS (2):
- vaccinated group (Experimental): evaluation of immunity's level against meningococcus C among people vaccinated in 2002 in Puy-de-Dôme
  Interventions: Other: Meningococcus C conjugate vaccine
- unvaccinate group (Other): Duration of vaccinal immunity, compare vaccinal immunity to possible natural immunity among unvaccinated people
  Interventions: Other: Meningococcus C conjugate vaccine

INTERVENTIONS:
Other: Meningococcus C conjugate vaccine

SUMMARY:
Meningococcus C vaccine was first used in France to prevent epidemics. It was a success in Puy-de-Dôme, Landes, Pyrénées Atlantiques and Hautes Pyrénées. Following many European countries, France introduced meningococcus C conjugate vaccine in 2009 but this recommendation was not suffiicently applied (6,6% of the 20-25 years-old were vaccinated in 2015).

The situation in France is very different from UK and there is no data on the subject. The vaccination campaign in 2002 in Puy-de-Dôme offers much more detachment, possible comparison between vaccinated and unvaccinated people, among which meningococcus circulation could maintain immunity. This is the reason why we have decided to assess in 2016 the vaccinal and natural immunity among Puy-de-Dôme population.

DETAILED DESCRIPTION:
People were recruited during hospitalisation or consultation of Pediatric, Occupational Medecine, Infectiology departments of Clermont Ferrand Hospital or Health Service of Auvergne's University, from March to September 2016.

Doctors gave informations about the study and collected consents before blood tests were done (two tubes of 4,5mL each).

Blood tests were daily collected and freezed. Then they were analysed at Meningococcus National Reference Center, in Paris.

ELIGIBILITY:
Inclusion Criteria:

* - people from 13 to 39 years old
* who received meningococcus C conjugate vaccine in 2002 in Puy-de-Dôme (vaccinated group) or not (unvaccinated group)

Exclusion Criteria:

* vaccination before or after 2002 containing meningococcus C valence
* refusal to participate

Ages: 13 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation in 2016 of immunity's level (antibodies) against meningococcus C among people vaccinated in 2002 in Puy-de-Dôme | at day 1

SECONDARY OUTCOMES:
Evaluate the duration (years) of vaccinal immunity | at day 1
Compare vaccinal immunity to possible natural immunity (antibodies level) among unvaccinated people | at day 1
Determine the cutt-off (age) for which vaccinal immunity is still protective (sufficient antibodies level) | at day 1
Adjust results on sociodemographic data (age, sex, city, number of years spent in Puy de Dôme, Auvergne, France and abroad from 2002 to 2016) | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean BEYTOUT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France